CLINICAL TRIAL: NCT01866943
Title: Role of Topical Tranexamic Acid in Total Hip Arthroplasty
Acronym: TXA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Jose Rodriguez, MD, Chieff Of Adult Reconstruction, Department of Orthopedics, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-253
Record Dates: First submitted 2013-05-29; First posted 2013-06-03 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-02

CONDITIONS: Post Operative Blood Loss
Keywords: Blood Loss; Tranexamic Acid; Total Hip Arthroplasty; Post Op; Post Operative; Prevent Post Operative Blood Loss
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1 (Placebo Comparator): Patients undergo primary total hip arthroplasty and have a wash of 100cc of normal saline applied to the tissues under the skin prior to skin closure. The wash sits in the wound for 5 minutes then is suctioned out and the skin is closed.
  Interventions: Drug: Normal Saline Solution
- Group 2 (Experimental): Patients undergo primary total hip arthroplasty and have a wash of 100cc of normal saline plus 1.5 g (100 mg/mL)Tranexamic Acid is applied to the tissues under the skin prior to skin closure. The wash sits in the wound for 5 minutes then is suctioned out and the skin is closed.
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — Tranexamic Acid 1.5 g (100 mg/mL)in 100cc normal saline is applied topically to the wound for 5 minutes time then suctioned and the skin closed. The control group receives just normal saline and no drug.
  Arms: Group 2
Drug: Normal Saline Solution
  Arms: Group 1

SUMMARY:
Total hip arthroplasty (THA) is a procedure associated with perioperative blood loss, requiring blood transfusions in some patients. The major cause of this blood loss is due to surgical trauma that induces the clotting cascade and fibrinolysis. Several previous studies and meta-analyses have shown that tranexamic acid is an effective antifibrinolytic agent that reduces blood loss in a variety of situations. Tranexamic acid given in an intravenous form has been extensively studied and shown to be efficacious in cardiothoracic, spine surgical procedures as well as total knee arthroplasty (TKA) and THA. Similarly, topical tranexamic acid has been associated with decreased blood loss in cardiac surgeries as well. Recently, results from a prospective randomized study on the topical use of tranexamic acid in total knee arthroplasty found it to be effective for reducing postoperative blood loss. Taking all of the above into consideration we have proposed a study to evaluate effects of topical application of tranexamic acid on postoperative blood loss and blood transfusion on patients undergoing total hip arthroplasty. The aim of this study is to evaluate the efficacy of the topical application of tranexamic acid on blood loss in patients undergoing a primary unilateral total hip arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age.
* Male or female.
* Degenerative joint disease of hip joint.
* Primary uncemented total hip arthroplasty.
* Willingness to participate in the study, follow up at regular intervals

Exclusion Criteria:

* Known allergy to tranexamic acid
* History of any acquired disturbances of color vision
* Preoperative anemia on basis of pre-operative lab work up (a hemoglobin value of <11 g/dL in females and <12 g/dL in males)
* History of previous myocardial infarction
* History of arterial or venous thromboembolic disease
* History of fibrinolytic disorders requiring intraoperative antifibrinolytic treatment, coagulopathy in the past and/or as identified by a preoperative platelet count of <150,000/mm3, an international normalized ratio of >1.5, or a prolonged partial thromboplastin time
* Pregnancy (h/o any missed menstrual periods in a women of reproductive age group)
* Breastfeeding
* Refusal of blood products
* Preoperative use of anticoagulant therapy within five days before surgery
* Medical issues that may pose complications for surgery and would disqualify patient for surgery regardless of clinical trial (e.g. renal and hepatic failure)
* Major comorbidities (e.g. severe ischemic heart disease )
* Severe pulmonary disease
* Preoperative blood donation
* Participation in another clinical trial involving pharmaceutical drugs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-11; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- North Shore Long Island Jewish Lenox Hill Hospital, New York, New York, United States

REFERENCES:
- [Background] Tsutsumimoto T, Shimogata M, Ohta H, Yui M, Yoda I, Misawa H. Tranexamic acid reduces perioperative blood loss in cervical laminoplasty: a prospective randomized study. Spine (Phila Pa 1976). 2011 Nov 1;36(23):1913-8. doi: 10.1097/BRS.0b013e3181fb3a42. PMID 21289587
- [Background] Elwatidy S, Jamjoom Z, Elgamal E, Zakaria A, Turkistani A, El-Dawlatly A. Efficacy and safety of prophylactic large dose of tranexamic acid in spine surgery: a prospective, randomized, double-blind, placebo-controlled study. Spine (Phila Pa 1976). 2008 Nov 15;33(24):2577-80. doi: 10.1097/BRS.0b013e318188b9c5. PMID 19011538
- [Background] Bednar DA, Bednar VA, Chaudhary A, Farrokhyar F. Tranexamic acid for hemostasis in the surgical treatment of metastatic tumors of the spine. Spine (Phila Pa 1976). 2006 Apr 15;31(8):954-7. doi: 10.1097/01.brs.0000209304.76581.c5. PMID 16622388
- [Background] Eubanks JD. Antifibrinolytics in major orthopaedic surgery. J Am Acad Orthop Surg. 2010 Mar;18(3):132-8. PMID 20190103
- [Background] Charoencholvanich K, Siriwattanasakul P. Tranexamic acid reduces blood loss and blood transfusion after TKA: a prospective randomized controlled trial. Clin Orthop Relat Res. 2011 Oct;469(10):2874-80. doi: 10.1007/s11999-011-1874-2. Epub 2011 Apr 22. PMID 21512813
- [Background] Ishida K, Tsumura N, Kitagawa A, Hamamura S, Fukuda K, Dogaki Y, Kubo S, Matsumoto T, Matsushita T, Chin T, Iguchi T, Kurosaka M, Kuroda R. Intra-articular injection of tranexamic acid reduces not only blood loss but also knee joint swelling after total knee arthroplasty. Int Orthop. 2011 Nov;35(11):1639-45. doi: 10.1007/s00264-010-1205-3. Epub 2011 Jan 21. PMID 21253725
- [Background] Johansson T, Pettersson LG, Lisander B. Tranexamic acid in total hip arthroplasty saves blood and money: a randomized, double-blind study in 100 patients. Acta Orthop. 2005 Jun;76(3):314-9. PMID 16156456
- [Background] Molloy DO, Archbold HA, Ogonda L, McConway J, Wilson RK, Beverland DE. Comparison of topical fibrin spray and tranexamic acid on blood loss after total knee replacement: a prospective, randomised controlled trial. J Bone Joint Surg Br. 2007 Mar;89(3):306-9. doi: 10.1302/0301-620X.89B3.17565. PMID 17356139
- [Background] Niskanen RO, Korkala OL. Tranexamic acid reduces blood loss in cemented hip arthroplasty: a randomized, double-blind study of 39 patients with osteoarthritis. Acta Orthop. 2005 Dec;76(6):829-32. doi: 10.1080/17453670510045444. PMID 16470437
- [Background] Rajesparan K, Biant LC, Ahmad M, Field RE. The effect of an intravenous bolus of tranexamic acid on blood loss in total hip replacement. J Bone Joint Surg Br. 2009 Jun;91(6):776-83. doi: 10.1302/0301-620X.91B6.22393. PMID 19483232
- [Background] Abrishami A, Chung F, Wong J. Topical application of antifibrinolytic drugs for on-pump cardiac surgery: a systematic review and meta-analysis. Can J Anaesth. 2009 Mar;56(3):202-12. doi: 10.1007/s12630-008-9038-x. Epub 2009 Feb 12. PMID 19247741
- [Background] Abul-Azm A, Abdullah KM. Effect of topical tranexamic acid in open heart surgery. Eur J Anaesthesiol. 2006 May;23(5):380-4. doi: 10.1017/S0265021505001894. Epub 2006 Jan 27. PMID 16438759
- [Background] De Bonis M, Cavaliere F, Alessandrini F, Lapenna E, Santarelli F, Moscato U, Schiavello R, Possati GF. Topical use of tranexamic acid in coronary artery bypass operations: a double-blind, prospective, randomized, placebo-controlled study. J Thorac Cardiovasc Surg. 2000 Mar;119(3):575-80. doi: 10.1016/s0022-5223(00)70139-5. PMID 10694619
- [Background] Fawzy H, Elmistekawy E, Bonneau D, Latter D, Errett L. Can local application of Tranexamic acid reduce post-coronary bypass surgery blood loss? A randomized controlled trial. J Cardiothorac Surg. 2009 Jun 18;4:25. doi: 10.1186/1749-8090-4-25. PMID 19538741
- [Background] Hanif M, Nourei SM, Dunning J. Does the use of topical tranexamic acid in cardiac surgery reduce the incidence of post-operative mediastinal bleeding? Interact Cardiovasc Thorac Surg. 2004 Dec;3(4):603-5. doi: 10.1016/j.icvts.2004.07.005. PMID 17670322
- [Background] Wong J, Abrishami A, El Beheiry H, Mahomed NN, Roderick Davey J, Gandhi R, Syed KA, Muhammad Ovais Hasan S, De Silva Y, Chung F. Topical application of tranexamic acid reduces postoperative blood loss in total knee arthroplasty: a randomized, controlled trial. J Bone Joint Surg Am. 2010 Nov 3;92(15):2503-13. doi: 10.2106/JBJS.I.01518. PMID 21048170
- [Background] Sukeik M, Alshryda S, Haddad FS, Mason JM. Systematic review and meta-analysis of the use of tranexamic acid in total hip replacement. J Bone Joint Surg Br. 2011 Jan;93(1):39-46. doi: 10.1302/0301-620X.93B1.24984. PMID 21196541
- [Background] Zufferey P, Merquiol F, Laporte S, Decousus H, Mismetti P, Auboyer C, Samama CM, Molliex S. Do antifibrinolytics reduce allogeneic blood transfusion in orthopedic surgery? Anesthesiology. 2006 Nov;105(5):1034-46. doi: 10.1097/00000542-200611000-00026. PMID 17065899

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Patients undergo primary total hip arthroplasty and have a wash of 100cc of normal saline applied to the tissues under the skin prior to skin closure. The wash sits in the wound for 5 minutes then is suctioned out and the skin is closed.
  Normal Saline Solution
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 19 | 22
Completed | 0 (Unknown - the only spreadsheet available is de-identified and blinded.) | 0 (Unknown - the only spreadsheet available is de-identified and blinded.)
Not Completed | 19 | 22

BASELINE CHARACTERISTICS:
Population: Baseline population to receive THA and be randomized to either Group 1 or Group 2.
Groups:
- All Study Participants: Baseline population, Groups are as follows:
  Group 1 (Normal Saline Solution) Patients undergo primary total hip arthroplasty and have a wash of 100cc of normal saline applied to the tissues under the skin prior to skin closure. The wash sits in the wound for 5 minutes then is suctioned out and the skin is closed.
  Group 2 (Tranexamic Acid) Patients undergo primary total hip arthroplasty and have a wash of 100cc of normal saline plus 1.5 g (100 mg/mL)Tranexamic Acid is applied to the tissues under the skin prior to skin closure. The wash sits in the wound for 5 minutes then is suctioned out and the skin is closed.
  Tranexamic Acid: Tranexamic Acid 1.5 g (100 mg/mL)in 100cc normal saline is applied topically to the wound for 5 minutes time then suctioned and the skin closed. The control group receives just normal saline and no drug.
  Since only blinded and deidentified data is available, Baseline measures will be reported on the entire population.
Arm/Group | All Study Participants
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants] — Population: Data are only available for the population overall since data were blinded and de-identified and it is not possible to determine what study subjects belong to which group. Further, since the study was terminated, no analysis was performed.
  Participants
    <=18 years | 0
    Between 18 and 65 years | 29
    >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.6 (9.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 19

OUTCOME MEASURES:

1. Primary Outcome: Estimated Blood Loss
Description: Estimated Blood Loss defined as Pre Op Hgb mins the Post Op Day two Hgb.
Time Frame: Pre Op, Post Op Day 2
Population: Patients undergoing primary unilateral THA. Group membership is unknown as only data available is blinded and de-identified.
Measure: Mean (Standard Deviation); unit: Hemoglobin (grams/deciliter)
Groups:
- Baseline Population: Data for 12 subjects is available, and cannot determine between groups as only data available is de-identified and blinded. Reporting data for these 12 subjects.
Arm/Group | Baseline Population
Number analyzed (Participants) | 12
Hemoglobin (grams/deciliter) | 2.93 (.77)

2. Secondary Outcome: Mid Thigh Circumference
Description: Measurement of the thigh at the half way point between the prominence of the greater trochanter and the lateral epicondyle of the femur. No data recorded at 2 weeks or 6 weeks for this study population.
Time Frame: Pre Op
Population: Patients undergoing primary unilateral THA.
Measure: Mean (Standard Deviation); unit: centimeters
Groups:
- Baseline Population: Data for this outcome measure is available for 16 subjects, and cannot determine between groups as only data available is de-identified and blinded. Therefore data for these 16 subjects is reported.
Arm/Group | Baseline Population
Number analyzed (Participants) | 16
centimeters | 52.99 (6.32)

3. Secondary Outcome: Harris Hip Scores
Description: Standardized questionnaire that measures clinical function related to the hip. Total potential range is from 4.0 - 96.0. A higher score indicates a more favorable clinical outcome.
Time Frame: Preoperative
Population: Patients undergoing primary total hip arthroplasty.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- All Study Participants: Data for this outcome is available for 4 subjects, and group membership is unknown as all data available is de-identified and blinded. Therefore data in these 4 subjects is reported.
Arm/Group | All Study Participants
Number analyzed (Participants) | 4
units on a scale | 58.34 (17.66)

4. Secondary Outcome: Harris Hip Scores
Description: as for outcome 3
Time Frame: 2 week
Population: Patients undergoing primary total hip arthroplasty.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- All Study Participants: Data for this outcome is available for 35 subjects, and group membership is unknown as all data available is de-identified and blinded. Therefore data in these 35 subjects is reported.
Arm/Group | All Study Participants
Number analyzed (Participants) | 35
units on a scale | 65.76 (20.80)

5. Secondary Outcome: Harris Hip Scores
Description: as for outcome 3
Time Frame: 6 week
Population: Patients undergoing primary total hip arthroplasty.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- All Study Participants: Data for this outcome is available for 31 subjects, and group membership is unknown as all data available is de-identified and blinded. Therefore data in these 31 subjects is reported.
Arm/Group | All Study Participants
Number analyzed (Participants) | 31
units on a scale | 81.77 (16.28)

ADVERSE EVENTS:
Time Frame: 6 weeks.
Description: Patients will be monitored every day until discharge from the hospital for any serious or other adverse events.
  Routine follow up will be done post-operatively at least up to one year to monitor any serious or other possible adverse events. Patients follow up at 3 months and 1 year post-surgery.
  Unblinding will be carried out only in the scenario of a serious adverse event (SAE) for the respective patient/s, with the help of research pharmacist maintaining the randomization record.
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/22
Other Adverse Events (participants affected / at risk) | 0/19 | 0/22

LIMITATIONS AND CAVEATS:
The study team is limited by a change in personnel. The data is not available classified by group: the only spreadsheet is incomplete, blinded and de-identified. The previous personnel have been contacted and are not cooperative.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No